CLINICAL TRIAL: NCT04108039
Title: Suppression of Endogenous Luteinizing Hormone (LH) Surge With Progesterone vs GnRH Antagonist in Freeze-all IVF Cycles. A Prospective Equivalence Study With Repeated Ovarian Stimulation Cycles.
Brief Title: Micronized Progesterone vs Gonadotropin-releasing Hormone (GnRH) Antagonist in Freeze-all IVF Cycles.
Acronym: Prog_STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Nikolaos Polyzos, Clinical and Scientific Director of Dexeus Mujer, Fundacion Dexeus
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FSD-PRG-2019-02
Record Dates: First submitted 2019-09-20; First posted 2019-09-27 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Infertility; IVF; Preimplantation Diagnosis
MeSH Terms: conditions — Infertility | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix; ganirelix; Progesterone; Utrogestan

STUDY DESIGN:
Intervention Model Description: 44 women undergoing IVF treatments due to infertility, will be asked to participate in a trial in which they will undergo 2 ovarian stimulation protocols with recombinant follicle stimulating hormone (rFSH): the first one using a flexible antagonist protocol to suppress the endogenous LH rise and the second using oral micronized progesterone 200 mg/day from day 1 of stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRH antagonist (Active Comparator): In the antagonist cycle, LH suppression will be accomplished by subcutaneous (SC) injections of 0.25 mg of Cetrorelix or Ganirelix starting in the presence of follicles >14mm or E2 levels >400 pg/ml and continuing until ovulation triggering.
  Interventions: Drug: GnRh antagonist
- Micronized progesterone (Experimental): In the progesterone cycle, endogenous LH suppression will be accomplished by oral administration of micronized progesterone (200 mg) once a day at bed time, from stimulation day 1 and continuing until ovulation triggering.
  Interventions: Drug: Micronized progesterone

INTERVENTIONS:
Drug: GnRh antagonist — In the antagonist cycle, LH suppression will be accomplished by subcutaneous (SC) injections of 0.25 mg of Cetrorelix or Ganirelix starting in the presence of follicles >14mm or E2 levels >400 pg/ml and continuing until ovulation triggering to avoid LH surge in COS
  Other Names: Cetrorelix or Ganirelix
  Arms: GnRH antagonist
Drug: Micronized progesterone — Micronized progesterone protocol to avoid LH surge in COS, from stimulation day 1 and continuing until ovulation triggering.
  Other Names: Utrogestan
  Arms: Micronized progesterone

SUMMARY:
To examine whether the number of euploid embryos following ovarian stimulation with micronized progesterone is equivalent as compared with the number of embryos after ovarian stimulation with the use of a GnRH antagonist in patients undergoing ovarian stimulation for IVF or intracytoplasmatic sperm injection (ICSI).

DETAILED DESCRIPTION:
The pre-ovulatory surges of GnRH and LH are activated by increased concentrations of circulating estradiol, but ovulation is blocked when progesterone concentrations are elevated, due to a central inhibition of the GnRH surge. Although traditionally GnRH has been traditionally considered the drug of choice to control endogenous LH in controlled ovarian stimulation (COS) cycles, recently, micronized progesterone has been shown to be an effective oral alternative for preventing premature LH surges during COS in women undergoing IVF/ICSI treatments, with excellent results, whereas their safety during pregnancy is well-established. This novel protocol, has several advantages (good tolerance, user convenience, and cost reduction), that are very attractive when it comes to establishing a convenient user regimen in combination with a ''freeze all'' strategy. However, the comparative efficacy of this novel protocol with the more universal use of GnRH-antagonist protocol for the treatment of IVF patients in terms of embryo ploidy has never been evaluated up to date. The current study aims, for the first time, to examine whether the number of euploid embryos following ovarian stimulation with micronized progesterone is equivalent as compared with the number of embryos after ovarian stimulation with the use of a GnRH antagonist in patients undergoing ovarian stimulation for IVF/ICSI.

If efficacy would prove to be similar, with no impact on the chromosomal constitution of embryos, there will be obvious advantages for the preferential use of micronized progesterone over the antagonist protocol: oral administration is preferred over subcutaneous injection, and total cost of medication would be lower. This would be particularly interesting for the future in all "freeze all" protocols such as women undergoing ovarian stimulation for fertility preservation, preimplantation genetic screening and oocyte donation programs.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients
* Age 36-40 years old
* BMI 18-30 kg/m2
* Undergoing preimplantation genetic screening cycles
* Planned to undergo at least two treatment cycles, to accumulate embryos to increase the chance of obtaining euploid embryos for transfer
* Willing to participate in the study

Exclusion Criteria:

* Age> 41
* Severe male factor requiring TESE (testicular sperm extraction)
* Low ovarian reserve (AMH < 1.2 ng/ml)
* Administration of any other drug potentially interfering with the treatment.

Ages: 36 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Number of euploid embryos as compared between the 2 ovarian stimulation cycles | 15-45 days following oocyte retrieval procedure
  Number of euploid embryos between oocytes received from the antagonist GnRh protocol or the micronized progesterone protocol.

SECONDARY OUTCOMES:
Endocrine profile at specific intervals | Stimulation day 0, day 6, day 8, day of final oocyte maturation and day +1 after oocyte maturation (actual day may vary between 9-15)
  To evaluate the difference in the mean serum estradiol (E2) levels (measured in pg/mL) at the predefined intervals treatment days.
Endocrine profile at specific intervals | Stimulation day 0, day 6, day 8, day of final oocyte maturation and day +1 after oocyte maturation (actual day may vary between 9-15)
  To evaluate the difference in the mean serum follicle stimulating hormone levels (FSH, measured in IU/mL) at the predefined intervals treatment days.
Endocrine profile at specific intervals | Stimulation day 0, day 6, day 8, day of final oocyte maturation and day +1 after oocyte maturation (actual day may vary between 9-15)
  To evaluate the difference in the mean serum progesterone levels (measured in ng/mL) at the predefined intervals treatment days.
Duration of stimulation | 9-20 days from initiation of ovarian stimulation
  Total days of ovarian stimulation. The outcome will be evaluated on the of final oocyte maturation.
Incidence of premature LH rise | 9-20 days from initiation of ovarian stimulation
Total dose of gonadotropins | 9-20 days from initiation of ovarian stimulation
  Total units of recombinant FSH. The outcome will be evaluated on the day of final oocyte maturation.
Number of mature oocytes | 9-20 days from initiation of ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Ultrasound ovarian follicles diameter measurement | 9-20 days from initiation of ovarian stimulation
  During the regular follicular scan, two diameters of each ovarian follicle will be recorded: the maximum diameters in the transverse and longitudinal scan planes.
Fertilization rate | 1 day after oocyte retrieval
  The outcome will be evaluated the day after the of oocyte retrieval

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitari Dexeus, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Mao X, Wang Y, Chen Q, Lu X, Hong Q, Kuang Y. Neonatal outcomes and congenital malformations in children born after human menopausal gonadotropin and medroxyprogesterone acetate treatment cycles. Arch Gynecol Obstet. 2017 Dec;296(6):1207-1217. doi: 10.1007/s00404-017-4537-z. Epub 2017 Sep 25. PMID 28948397
- [Background] Zhu X, Ye H, Fu Y. Use of Utrogestan during controlled ovarian hyperstimulation in normally ovulating women undergoing in vitro fertilization or intracytoplasmic sperm injection treatments in combination with a "freeze all" strategy: a randomized controlled dose-finding study of 100 mg versus 200 mg. Fertil Steril. 2017 Feb;107(2):379-386.e4. doi: 10.1016/j.fertnstert.2016.10.030. Epub 2016 Nov 16. PMID 27865446
- [Background] Zhu X, Zhang X, Fu Y. Utrogestan as an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Medicine (Baltimore). 2015 May;94(21):e909. doi: 10.1097/MD.0000000000000909. PMID 26020402
- [Background] Lambalk CB, Banga FR, Huirne JA, Toftager M, Pinborg A, Homburg R, van der Veen F, van Wely M. GnRH antagonist versus long agonist protocols in IVF: a systematic review and meta-analysis accounting for patient type. Hum Reprod Update. 2017 Sep 1;23(5):560-579. doi: 10.1093/humupd/dmx017. PMID 28903472
- [Background] Verberg MF, Eijkemans MJ, Heijnen EM, Broekmans FJ, de Klerk C, Fauser BC, Macklon NS. Why do couples drop-out from IVF treatment? A prospective cohort study. Hum Reprod. 2008 Sep;23(9):2050-5. doi: 10.1093/humrep/den219. Epub 2008 Jun 10. PMID 18544578
- [Background] Richter TA, Robinson JE, Lozano JM, Evans NP. Progesterone can block the preovulatory gonadotropin-releasing hormone/luteinising hormone surge in the ewe by a direct inhibitory action on oestradiol-responsive cells within the hypothalamus. J Neuroendocrinol. 2005 Mar;17(3):161-9. doi: 10.1111/j.1365-2826.2005.01287.x. PMID 15796768
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Griesinger G, Venetis CA, Tarlatzis B, Kolibianakis EM. To pill or not to pill in GnRH-antagonist cycles: the answer is in the data already! Reprod Biomed Online. 2015 Jul;31(1):6-8. doi: 10.1016/j.rbmo.2015.04.001. Epub 2015 Apr 9. PMID 25985996
- [Background] Devroey P, Polyzos NP, Blockeel C. An OHSS-Free Clinic by segmentation of IVF treatment. Hum Reprod. 2011 Oct;26(10):2593-7. doi: 10.1093/humrep/der251. Epub 2011 Aug 9. PMID 21828116
- [Background] Cedrin-Durnerin I, Bstandig B, Parneix I, Bied-Damon V, Avril C, Decanter C, Hugues JN. Effects of oral contraceptive, synthetic progestogen or natural estrogen pre-treatments on the hormonal profile and the antral follicle cohort before GnRH antagonist protocol. Hum Reprod. 2007 Jan;22(1):109-16. doi: 10.1093/humrep/del340. Epub 2006 Aug 26. PMID 16936304
- [Background] Dong J, Wang Y, Chai WR, Hong QQ, Wang NL, Sun LH, Long H, Wang L, Tian H, Lyu QF, Lu XF, Chen QJ, Kuang YP. The pregnancy outcome of progestin-primed ovarian stimulation using 4 versus 10 mg of medroxyprogesterone acetate per day in infertile women undergoing in vitro fertilisation: a randomised controlled trial. BJOG. 2017 Jun;124(7):1048-1055. doi: 10.1111/1471-0528.14622. PMID 28276192
- [Derived] Vidal MDM, Martinez F, Rodriguez I, Polyzos NP. Ovarian response and embryo ploidy following oral micronized progesterone-primed ovarian stimulation versus GnRH antagonist protocol. A prospective study with repeated ovarian stimulation cycles. Hum Reprod. 2024 May 2;39(5):1098-1104. doi: 10.1093/humrep/deae047. PMID 38498835